CLINICAL TRIAL: NCT04406623
Title: Phase 1 Dose Escalation Study of the Agonist Redirected Checkpoint, SL-172154 (SIRPα-Fc-CD40L) Administered Intravenously in Subjects With Ovarian Cancer
Brief Title: Phase 1 Study of SL-172154 (SIRPα-Fc-CD40L) in Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shattuck Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SL03-OHD-101
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SL-172154 (Experimental): Intravenous administration
  Interventions: Drug: SL-172154

INTERVENTIONS:
Drug: SL-172154 — The investigational product (IP), SL-172154, is a novel fusion protein consisting of human SIRPα and CD40L (SIRPα -Fc-CD40L) linked via a human Fc.

SUMMARY:
This is a Phase 1 first in human, open label, multi-center, dose escalation study to evaluate the safety, tolerability, PK, anti-tumor activity and pharmacodynamic effects of SL-172154 in subjects with ovarian cancer.

DETAILED DESCRIPTION:
This Phase 1 trial will evaluate the safety, tolerability, pharmacokinetics, anti-tumor and pharmacodynamic effects of SL-172154 and identify the dose and schedule i.e., recommended Phase 2 dose for future development (RP2D). Subjects eligible for enrollment are required to have platinum-ineligible ovarian, fallopian tube, and primary peritoneal cancers. The study design consists of dose escalation cohorts, an optional pharmacodynamic cohort, and an optional dose expansion cohort. In the dose escalation phase of the study, subjects will be enrolled into sequential dose levels. The study may also enroll a pharmacodynamic cohort to obtain additional pharmacodynamic data at one or more dose levels that have completed evaluation for safety without exceeding the maximum tolerated dose (MTD). Subjects enrolled in the pharmacodynamic cohort will not inform dose escalation decisions. A dose expansion cohort may be opened to further characterize safety, tolerability, PK, anti-tumor activity, and pharmacodynamic data to inform the selection of a RP2D.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. Subject has voluntarily agreed to participate by giving written informed consent in accordance with ICH/GCP guidelines and applicable local regulations.
2. Subject must have a histologically confirmed diagnosis of an unresectable, locally advanced or metastatic ovarian cancer, or primary peritoneal cancer or fallopian tube cancer.
3. Subjects must be refractory or intolerant to existing therapy(ies) known to provide clinical benefit for their condition. Subject must have received platinum-based therapies, and should not be eligible for further platinum therapy, or should be intolerant to such therapy. Subjects with HRD positive disease may participate if they have received prior polyadenosine diphosphate ribose polymerase (PARP) inhibitor therapy given alone or with bevacizumab.
4. Subjects should not be primary platinum refractory as defined by progressing during or within 1 month of upfront platinum therapy.
5. Has measurable disease by RECIST v1.1 using radiologic assessment.
6. Subject age is 18 years and older.
7. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
8. Has life expectancy of greater than 12 weeks.
9. Has adequate organ function.
10. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 72 hours of D1 of IP.
11. Recovery from prior anti-cancer treatments including surgery, radiotherapy, chemotherapy or any other anti-cancer therapy to baseline or ≤ Grade 1.
12. Willing to consent to mandatory pre-treatment and on-treatment tumor biopsy(ies), unless there is excessive risk as determined by the investigator.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Prior treatment with an anti-CD47 or anti-SIRPα targeting agent or a CD40 agonist.
2. Any anti-cancer therapy within the washout period prior to first dose (D1) of SL-172154.
3. Concurrent chemotherapy, immunotherapy, biologic or hormonal/hormonal suppression therapy for cancer treatment is prohibited. Concurrent use of hormones for non-cancer related conditions is acceptable.
4. Use of corticosteroids or other immunosuppressive medication, current or within 14 days of D1 of SL-172154 treatment.
5. Receipt of live attenuated vaccine within 28 days of D1 of IP.
6. Active or documented history of autoimmune disease. Exceptions include controlled Type I diabetes, vitiligo, alopecia areata or hypo/hyperthyroidism.
7. Hypersensitivity to the active drug substance or to any of the excipients for the agent to be administered or subjects with known hypersensitivity to Chinese hamster ovary cell products.
8. Active pneumonitis (i.e. drug-induced, idiopathic pulmonary fibrosis, radiation-induced, etc.).
9. Ongoing or active infection (e.g., no systemic antimicrobial therapy for treatment of infection within 5 days of D1 of IP).
10. Symptomatic peptic ulcer disease or gastritis, active diverticulitis, other serious gastrointestinal disease associated with diarrhea within 6 months of D1 of IP.
11. Clinically significant or uncontrolled cardiac/thromboembolic disease.
12. Untreated central nervous system or leptomeningeal metastases.
13. Women who are breast feeding.
14. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or compromised ability to provide written informed consent.
15. Another malignancy that requires active therapy and that in the opinion of the investigator and Sponsor would interfere with monitoring of radiologic assessments of response to IP.
16. Has undergone allogeneic stem cell transplantation or organ transplantation.
17. Known history or positive test for human immunodeficiency virus, or positive test for hepatitis B.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - START Midwest, Grand Rapids, Michigan
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Stephenson Cancer Center at Oklahoma University, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - START Mountain Region, West Valley City, Utah

REFERENCES:
- [Derived] Lakhani NJ, Stewart D, Richardson DL, Dockery LE, Van Le L, Call J, Rangwala F, Wang G, Ma B, Metenou S, Huguet J, Offman E, Pandite L, Hamilton E. First-in-human phase I trial of the bispecific CD47 inhibitor and CD40 agonist Fc-fusion protein, SL-172154 in patients with platinum-resistant ovarian cancer. J Immunother Cancer. 2025 Jan 11;13(1):e010565. doi: 10.1136/jitc-2024-010565. PMID 39800375

RESULTS

PARTICIPANT FLOW:
Groups:
- SL-172154 (0.1 mg/kg): 0.1 mg/kg of SL-172154 (Schedule 1)
- SL-172154 (0.3 mg/kg): 0.3 mg/kg of SL-172154 (Schedule 1 or Schedule 2)
- SL-172154 (1.0 mg/kg): 1.0 mg/kg of SL-172154 (Schedule 1)
- SL-172154 (3.0 mg/kg): 3.0 mg/kg of SL-172154 (Schedule 1 or Schedule 2)
- SL-172154 (10.0 mg/kg): 10.0 mg/kg of SL-172154 (Schedule 1)
Period: Overall Study
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Started | 3 | 6 | 4 | 9 | 5
Completed | 3 | 6 | 4 | 9 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SL-172154 (0.1 mg/kg): 0.1 mg/kg of IV SL-172154 (Schedule 1)
- SL-172154 (0.3 mg/kg): 0.3 mg/kg of IV SL-172154 (Schedule 1 or Schedule 2)
- SL-172154 (1.0 mg/kg): 1.0 mg/kg of IV SL-172154 (Schedule 1)
- SL-172154 (3.0 mg/kg): 3.0 mg/kg of IV SL-172154 (Schedule 1 or Schedule 2)
- SL-172154 (10.0 mg/kg): 10.0 mg/kg of IV SL-172154 (Schedule 1)
- Total: Total of all reporting groups
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg) | Total
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5 | 27
Age, Continuous [Median (Full Range); unit: years] | 72.0 [71 to 77] | 65.0 [33 to 70] | 60.5 [47 to 64] | 68.0 [59 to 85] | 67.0 [52 to 76] | 66.0 [33 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 9 | 5 | 27
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 2 | 9 | 5 | 24
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 3
  White | 2 | 6 | 2 | 8 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of SL-172154
Description: Number of participants with treatment emergent adverse events
Time Frame: From Day 1 to 90 days after Last Dose of SL-172154
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
Participants | 3 | 6 | 4 | 9 | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD) of SL-172154
Description: Number of participants with dose limiting toxicities (DLTs)
Time Frame: From Day 1 to 90 days after Last Dose of SL-172154
Population: DLT evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 5
Participants | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Recommended Phase 2 Dose (RP2D) for SL-172154
Description: Based on review of all data, including safety, tolerability, PK, antitumor activity, and PD effects
Time Frame: Approximately 24 months
Measure: Number; unit: mg/kg
Groups:
- SL-172154: Schedule 1: IV SL-172154 given on Days 1, 8, and 15 of Cycle 1 (28 days) and Days 1 and 15 of all additional cycles (28 days each)
Arm/Group | SL-172154
Number analyzed (Participants) | 27
mg/kg | 3.0

4. Secondary Outcome: Assess Preliminary Evidence of Anti-tumor Activity of SL-172154
Description: Number of participants with an objective response per investigator assessment according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1). Objective response includes complete response (disappearance of all target lesions) and partial response (>/= 30% decrease in the sum of the longest diameter of target lesions).
Time Frame: Approximately 24 months
Population: Response Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Immunogenicity to SL-172154
Description: Number of participants with positive anti-drug antibody (ADA) titer, sustained ADA response (positive ADA in >/= 2 samples without reverting to negative ADA or positive ADA in the last sample), or persistent ADA response (positive ADA in >/= 2 samples where the first and last samples are >/= 16 weeks apart, or positive ADA in the last sample, or only one sample but < 16 weeks before a negative last sample).
Time Frame: Approximately 24 months
Population: Immunogenicity Population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
Participants
  Positive anti-drug antibody titer | 1 | 4 | 2 | 3 | 3
  Sustained ADA response | 1 | 3 | 2 | 1 | 1
  Persistent ADA response | 0 | 1 | 1 | 1 | 0

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of SL-172154
Description: The Cmax is the maximum observed serum concentration of SL-172154 following single and multiple doses
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
ng/mL
  Cycle 1 Day 1 | 117.68 (31.06) | 126.33 (89.20) | 545.03 (406.44) | 4593.19 (90.34) | 87509.31 (51.12)
  Cycle 1 Day 15 | 59.20 (29.92) | 136.96 (93.93) | 1772.77 (111.10) | 3071.26 (883.11) | 50484.31 (33.38)
  Cycle 2 Day 1 | 72.96 (55.09) | 82.11 (14.84) | 1240.25 (72.61) | 5219.40 (151.02) | 115536.25 (51.83)

7. Secondary Outcome: Minimum Serum Concentration (Cmin) of SL-172154
Description: The Cmin is the minimum observed serum concentration of SL-172154 following at least one dose
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1 (each cycle = 28 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 3 | 8 | 3
ng/mL
  Cycle 1 Day 15 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0
  Cycle 2 Day 1 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0 | 0 (NA) — Coefficient of variation cannot be determined when mean is 0

8. Secondary Outcome: Time at Which Maximum Concentration of SL-172154 is Observed (Tmax)
Description: The Tmax is the time at which the maximum concentration of SL-172154 is observed following single and multiple doses
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
hours
  Cycle 1 Day 1 | 0.5 [0.5 to 0.5] | 0.56 [0.5 to 1.6] | 0.55 [0.5 to 2.6] | 2.53 [1.1 to 5.0] | 3.43 [2.0 to 5.0]
  Cycle 1 Day 15 | 0.53 [0.5 to 0.7] | 0.54 [0.5 to 2.3] | 0.57 [0.5 to 0.6] | 2.06 [1.1 to 2.8] | 3.6 [2.0 to 3.6]
  Cycle 2 Day 1 | 0.5 [0.5 to 0.5] | 0.53 [0.5 to 1.1] | 0.55 [0.5 to 1.5] | 2.08 [1.0 to 4.1] | 1.97 [1.9 to 2.0]

9. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC)
Description: The AUC is the area under the serum concentration time curve following single and multiple doses of SL-172154. AUC (0-last; from time 0 to the last quantifiable concentration) is reported for C1D1 and AUC (tau; over a dosing interval) is reported for C1D15 and C2D1.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
hours*ng/mL
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 143.54 (7.74) | 639.40 (18.47) | 7062.14 (81.59) | 200095.11 (78.74)
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 13030.1 (27.31) | 133015.0 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification
  Cycle 2 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 6103.60 (130.09) | 236849.02 (91.90)

10. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life (t1/2) of SL-172154
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
hours
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.50 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.37 (0.056) | 0.75 (0.710) | 0.86 (0.278)
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.32 (0.132) | 0.71 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification
  Cycle 2 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.36 (0.158) | 1.30 (0.477)

11. Secondary Outcome: Clearance (CL)
Description: Clearance of SL-172154
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
liters per hour
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 110.64 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 121.22 (46.305) | 35.73 (25.580) | 4.13 (2.605)
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 15.15 (2.650) | 4.44 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification
  Cycle 2 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 44.88 (48.958) | 3.17 (1.637)

12. Secondary Outcome: Volume of Distribution
Description: Volume of distribution of SL-172154
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 5
liters
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 79.83 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 64.28 (28.528) | 28.46 (17.148) | 4.84 (2.982)
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 7.32 (4.187) | 4.53 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification
  Cycle 2 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 32.01 (49.282) | 5.62 (3.337)

ADVERSE EVENTS:
Time Frame: Subjects were followed continuously for all AEs starting when a subject signed the informed consent form, throughout the course of treatment, and for 90 days after the last dose of study treatment, an average of 10.5 weeks.
Arm/Group | SL-172154 (0.1 mg/kg) | SL-172154 (0.3 mg/kg) | SL-172154 (1.0 mg/kg) | SL-172154 (3.0 mg/kg) | SL-172154 (10.0 mg/kg)
All-Cause Mortality (participants affected / at risk) | 2/3 | 5/6 | 3/4 | 2/9 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 1/4 | 2/9 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL-172154 (0.1 mg/kg) (N=3) | SL-172154 (0.3 mg/kg) (N=6) | SL-172154 (1.0 mg/kg) (N=4) | SL-172154 (3.0 mg/kg) (N=9) | SL-172154 (10.0 mg/kg) (N=5)
embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SL-172154 (0.1 mg/kg) (N=3) | SL-172154 (0.3 mg/kg) (N=6) | SL-172154 (1.0 mg/kg) (N=4) | SL-172154 (3.0 mg/kg) (N=9) | SL-172154 (10.0 mg/kg) (N=5)
infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 8 | 5
nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 1
constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2
diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1
abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
fatigue (General disorders) | 3 | 4 | 1 | 2 | 2
chills (General disorders) | 0 | 0 | 1 | 1 | 1
pain (General disorders) | 0 | 1 | 0 | 1 | 1
oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1
dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
AST increased (Investigations) | 0 | 1 | 0 | 1 | 2
ALT increased (Investigations) | 0 | 1 | 0 | 1 | 1
activated PTT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1
blood LDH increased (Investigations) | 0 | 0 | 0 | 0 | 2
headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
pruritis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2
embolism (Vascular disorders) | 1 | 0 | 0 | 1 | 0
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site agrees not to publish any Study Results or data before the publication of results from the Overall Study. After Sponsor has published the results of the Overall Study, Site may publish or present results generated at Site. If Sponsor has not published results of the Overall Study within 18 months of data base lock, Site may publish the results of the Study that were generated at Site. Site agrees to first submit to Sponsor the proposed publication at least 30 days prior to the submission.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04406623/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT04406623/SAP_001.pdf